CLINICAL TRIAL: NCT04543526
Title: A Post-market Observational Study With the easyEndoTM Universal Linear Cutting Stapler in Standard Laparoscopic and Robot-assisted Laparoscopic Roux-en-Y Gastric Bypass (RYGB) Surgery
Acronym: SIRIUS
Status: Withdrawn | Type: Observational
Why Stopped: No CEC approval
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: DM-ZOL-01
Record Dates: First submitted 2020-08-13; First posted 2020-09-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients: Obese patients eligible for standard laparoscopic or robot-assisted laparoscopic RYGB surgery.
  Interventions: Device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical)

INTERVENTIONS:
Device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) — Investigational device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical). Device for creating anastomoses during standard and robot-assisted laparoscopic RYGB, manufactured by Ezisurg Medical.

SUMMARY:
The primary purpose of this observational registry is to evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads from Ezisurg Medical when used to create anastomoses during standard and robot-assisted laparoscopic Roux-en-Y Gastric Bypass (RYGB) surgery. Stapler performance during surgery as well as post-operative pain and the clinical efficacy of the procedures will be determined as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age at study entry.
* Patient and investigator signed and dated the informed consent form prior to the index-procedure.
* Patient has a BMI ≥ 35 kg/m2 with one or more related co-morbidity.
* Patient has a BMI ≥ 40 kg/m2.
* Patient is eligible for standard laparoscopic or for robotic-assisted laparoscopic RYGB surgery.

Exclusion Criteria:

* Patient is unable / unwilling to provide informed consent.
* Patient has a history of bariatric surgery.
* Patient is unable to comply with the study protocol or proposed follow-up visits.
* Patient has a contra-indication for standard laparoscopic or robot-assisted laparoscopic RYGB surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients eligible for standard laparoscopic or robot-assisted laparoscopic RYGB surgery. This registry will collect data from 150 laparoscopic RYGB procedures in which anastomoses are created with the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety - Conversion rate to laparotomy | At index procedure.
  Number of conversions to laparotomy during the index procedure
Safety - Length of stay at the intensive care unit | At index procedure.
  Number of days at the intensive care unit after the index procedure.
Safety - Length of stay in the hospital by the modified Post-Anesthesia Discharge Scoring System (PADSS) | At index procedure.
  The Modified PADSS guarantees safe discharge. PADSS is based on the assessment of 6 criteria: vital signs (including blood pressure, pulse, temperature and respiratory rate), ambulation, nausea / vomiting, pain, surgical bleeding and fluid intake / output. Each criterion is given a score from 0 to 2. Patients scoring ≥ 9 are considered fit for discharge, provided that the score for vital signs is not lower than 2 and that none of the other five criteria is 0, even if the total score reaches 9.
Safety - Number of re-interventions and number of participants with (serious) adverse events | At index procedure.
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety - Length of stay at the intensive care unit. | At discharge, up to 1 week.
  Number of days at the intensive care unit after the index procedure.
Safety - Length of stay in the hospital by the modified Post-Anesthesia Discharge Scoring System (PADSS) | At discharge, up to 1 week.
  he Modified PADSS guarantees safe discharge. PADSS is based on the assessment of 6 criteria: vital signs (including blood pressure, pulse, temperature and respiratory rate), ambulation, nausea / vomiting, pain, surgical bleeding and fluid intake / output. Each criterion is given a score from 0 to 2. Patients scoring ≥ 9 are considered fit for discharge, provided that the score for vital signs is not lower than 2 and that none of the other five criteria is 0, even if the total score reaches 9.
Safety - Number of re-interventions and number of participants with (serious) adverse events | At discharge, up to 1 week.
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety - Number of re-interventions and number of participants with (serious) adverse events | Follow-up 1: 1 month after the procedure.
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety - Number of re-interventions and number of participants with (serious) adverse events | Follow-up 2: 6 months after the procedure.
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety - Number of re-interventions and number of participants with (serious) adverse events | Follow-up 3: 12 months after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety - Number of re-interventions and number of participants with (serious) adverse events | Follow-up 4: 24 months after the procedure.
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.

SECONDARY OUTCOMES:
Device performance - Technical success of the surgical procedure performed with the device | At index procedure
  Number of procedures with technical success defined as bariatric surgery as intended, without technical difficulties and without conversion to laparotomy.
Device performance - Scoring of operator satisfaction | At index procedure
  Scoring of: easy of intra-abdominal device positioning, grasping/climbing force, sharpness of the blades, staple-line formation, device stability, device maneuverability, battery power, device consistency and reliability, ergonomic design, hemostasis. Each of the aforementioned items receives a score from 0 to 4, with 0 indicating that the user is very unsatisfied and 4 indicating that the user is very satisfied.
Post-operative pain by means of the Visual Analogue Scale (VAS) | At index procedure
  Assessment of acute post-operative abdominal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative pain by means of the Visual Analogue Scale (VAS) | At discharge, up to 1 week
  Assessment of acute post-operative abdominal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative pain by means of the Visual Analogue Scale (VAS) | Follow-up 1: 1 month after the procedure
  Assessment of the worst post-operative abdominal pain since discharge by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative food tolerance by means of the food tolerance questionnaire | Follow-up 1: 1 month after the procedure
  Food tolerance by means of the food tolerance questionnaire. The food tolerance questionnaire allows to score the patients' satisfaction regarding food intake and food tolerance after bariatric surgery. The patients' interpretation of food intake is scored between 1 (very poor) and 5 (excellent). A cumulative score, varying between 1 and 27 is derived, with 27 representing an excellent food tolerance.
Post-operative food tolerance by means of the food tolerance questionnaire | Follow-up 2: 6 months after the procedure
  Food tolerance by means of the food tolerance questionnaire. The food tolerance questionnaire allows to score the patients' satisfaction regarding food intake and food tolerance after bariatric surgery. The patients' interpretation of food intake is scored between 1 (very poor) and 5 (excellent). A cumulative score, varying between 1 and 27 is derived, with 27 representing an excellent food tolerance.
Post-operative food tolerance by means of the food tolerance questionnaire | Follow-up 3: 12 months after the procedure
  Food tolerance by means of the food tolerance questionnaire. The food tolerance questionnaire allows to score the patients' satisfaction regarding food intake and food tolerance after bariatric surgery. The patients' interpretation of food intake is scored between 1 (very poor) and 5 (excellent). A cumulative score, varying between 1 and 27 is derived, with 27 representing an excellent food tolerance.
Post-operative food tolerance by means of the food tolerance questionnaire | Follow-up 4: 24 months after the procedure
  Food tolerance by means of the food tolerance questionnaire. The food tolerance questionnaire allows to score the patients' satisfaction regarding food intake and food tolerance after bariatric surgery. The patients' interpretation of food intake is scored between 1 (very poor) and 5 (excellent). A cumulative score, varying between 1 and 27 is derived, with 27 representing an excellent food tolerance.
Post-operative change in weight | Follow-up 1: 1 month after the procedure
  Weight loss 1 month after the surgical procedure as compared to the patients' weight at baseline.
Post-operative change in weight | Follow-up 2: 6 months after the procedure
  Weight loss 6 months after the surgical procedure as compared to the patients' weight at baseline.
Post-operative change in weight | Follow-up 3: 12 months after the procedure
  Weight loss 12 months after the surgical procedure as compared to the patients' weight at baseline.
Post-operative change in weight | Follow-up 4: 24 months after the procedure
  Weight loss 24 months after the surgical procedure as compared to the patients' weight at baseline.
Number of participants with a post-operative change of cormorbidities | Follow-up 3: 12 months after the procedure
  Comorbidities (diabetes mellitus, peripheral arterial disease, coronary arterial disease, sleep disordered breathing, hypertension, dyslipidemia, hypercholesterolemia, hypertriglyceridemia, asthma, congestive heart failure, degenerative joint disease, gastroesophageal reflux, chronic obstructive pulmonary disease, use of immunosuppressants) 12 months after the surgical procedure as compared to the patients' comorbidities at baseline.
Number of participants with a post-operative change of cormorbidities | Follow-up 4: 24 months after the procedure
  Comorbidities (diabetes mellitus, peripheral arterial disease, coronary arterial disease, sleep disordered breathing, hypertension, dyslipidemia, hypercholesterolemia, hypertriglyceridemia, asthma, congestive heart failure, degenerative joint disease, gastroesophageal reflux, chronic obstructive pulmonary disease, use of immunosuppressants) 24 months after the surgical procedure as compared to the patients' comorbidities at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Verhelst, Dr., Principal Investigator — Ziekenhuis Oost-Limburg (ZOL)
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg (ZOL), Genk
  - Ziekenhuis Maas en Kempen (ZMK), Maaseik

IPD SHARING:
Plan to Share IPD: No